CLINICAL TRIAL: NCT01975025
Title: Hemodialysis Frequency and the Calcification Propensity of Serum
Acronym: Intensified HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 146/13
Record Dates: First submitted 2013-10-25; First posted 2013-11-04 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Hemodialysis; Anuria
Keywords: Renal Dialysis
MeSH Terms: conditions — Anuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All study participants (Experimental): Short daily dialysis for 2 weeks
  Interventions: Procedure: Short daily dialysis for 2 weeks

INTERVENTIONS:
Procedure: Short daily dialysis for 2 weeks

SUMMARY:
The aim of this clinical research project is to test the hypothesis that daily dialysis has favorable effects on the calcification propensity of human serum, when determined by the investigators' newly developed in vitro serum test. The investigators' hypothesis is that shorter interdialytic intervals will result in an improved calcification propensity of serum. The determination of serum calcification has the potential to become a novel measure of dialysis quality in the future.

DETAILED DESCRIPTION:
Background

The serum calcification test has been established and validated by A. Pasch and coworkers, the expertise to perform the necessary statistical analyses is present in the investigator's department, all patient-related procedures necessary for this project are routinely performed in the investigator's department.

Objective

Does short daily hemodialysis strengthen the calcification-inhibitory forces inherent in hemodialysis patient sera, when compared to conventional three-times weekly hemodialysis?

Methods

Serum calcification test

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemodialysis >3 months
* Anuria (<100ml urine per day)
* Written informed consent

Exclusion Criteria

* Citrate dialysis
* Significant fistula recirculation (>15%)
* Infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline calcification propensity of serum | 6 weeks

SECONDARY OUTCOMES:
Change from baseline of sodium, potassium, calcium, phosphate, magnesium, albumin, protein, hematocrit and their correlation with calcification propensity of serum | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Pasch, PD. Dr. med., Principal Investigator — University Clinic Inselspital Bern
Locations (1):
- Dep. of Nephrology, Hypertension and Clinical Pharmacology, Bern University Hospital, Bern, Canton of Bern, Switzerland